CLINICAL TRIAL: NCT00163657
Title: An Open-Label, Randomized, Prospective Multicenter Study To Compare The Efficacy And Safety Among 3 Immunosuppressant Treatment Regimens In Patients Receiving A Liver Transplant For ESLD Caused By Chronic Hepatitis C
Brief Title: Study of Liver Transplant For End-Stage Liver Disease Caused By Chronic Hepatitis C Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Baylor Health Care System (Other); Emory University (Other); University of Southern California (Other); Mayo Clinic - Scottsdale/Phoenix, Arizona (Unknown); New York Presbyterian Hospital (Other); Oregon Health and Science University (Other); New York University (Other); University of Cincinnati (Other); University of Alabama at Birmingham (Other); The University of Texas Health Science Center at San Antonio (Other); University of Chicago (Other); University of California, San Francisco (Other); Mayo Clinic - Rochester, Minnesota (Unknown); Medical University of South Carolina (Other); University of Virginia (Other); Lahey Clinic (Other); University of Medicine and Dentistry of New Jersey (Other); Northwestern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-01-L; ZEN159 (Other: Baylor Research Institute)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: End Stage Liver Disease; Hepatitis C
Keywords: Hepatitis C Virus; Immunosuppressive Agents
MeSH Terms: conditions — End Stage Liver Disease; Hepatitis C | interventions — Daclizumab; Tacrolimus; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- tacrolimus and cyclosporine (Active Comparator): immunosuppressant treatment regimens the intervention is antirejection treatment with the above labeled drugs tacrolimus and cyclosporine
  Interventions: Drug: Daclizumub; Drug: Tacrolimus
- MMF, tacrolimus and cyclosporine (Active Comparator): immunosuppressant treatment regimensthe intervention is antirejection treatment with the above labeled drugs MMF tacrolimus and cyclosporine
  Interventions: Drug: Tacrolimus; Drug: Cyclosporine; Drug: MMF
- daclizumub, MMFand tacrolimus (Active Comparator): immunosuppressant treatment regimens
  Interventions: Drug: Daclizumub; Drug: Tacrolimus; Drug: MMF

INTERVENTIONS:
Drug: Daclizumub — anti-rejection drug
  Other Names: Zenapax
  Arms: daclizumub, MMFand tacrolimus; tacrolimus and cyclosporine
Drug: Tacrolimus — anti rejection drug
  Other Names: Prograf
Drug: Cyclosporine — anti rejection drug
  Other Names: Neoral
  Arms: MMF, tacrolimus and cyclosporine
Drug: MMF — anti rejection drug
  Other Names: mycophenolate mofetil
  Arms: MMF, tacrolimus and cyclosporine; daclizumub, MMFand tacrolimus

SUMMARY:
The purpose of this study is to compare three treatment regimens in patients who have received a liver transplant for end-stage liver disease caused by Chronic Hepatitis C infection.

DETAILED DESCRIPTION:
End-stage liver disease due to Hepatitis C virus (HCV) infection is the most common reason for liver transplantation in the United States. Patients who have HCV will always carry the virus in their body. If patients respond to treatment, the virus is no longer active. This means that although the virus is still present, it is not currently causing damage to their liver.

Because recurrence of HCV is virtually universal in HCV positive transplant recipients and is associated with long term, possibly lethal complications, the search for the most appropriate therapies must also include methods to prevent or minimize recurrence or disease progression, if the goal of improving long term outcomes for these patients is to be achieved.

Corticosteroids and high doses of immunosuppressive agents have been associated with increased rates of HCV recurrence. Finding a regimen that provides adequate immunosuppression to prevent early and late rejection episodes, and minimizes steroid usage as well as high doses of other immunosuppressive agents is highly desirable.

This study is being conducted to determine the most effective immunosuppressive regimen that will prevent allograft rejection, minimize adverse events and at the same time, prevent or reduce the incidence of HCV recurrence following liver transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has been fully informed and has signed an IRB approved informed consent form and is willing and able to follow study procedures for the full 2 years.
2. Patient is a recipient of a primary whole/split, cadaveric/living donor liver transplant for end stage chronic Hepatitis C.
3. Patient is > age 18.
4. Female patients of child bearing potential must have a negative urine or serum pregnancy test upon hospitalization or within 7 days prior to enrollment and have agreed to utilize effective birth control throughout the study as well as for 6 weeks following study completion.

Exclusion Criteria:

1. Patient has previously received or is receiving an organ transplant other than a liver.
2. Patient has received a liver transplant from a Hepatitis B core antibody or a Hepatitis C antibody positive donor.
3. Patient has received an ABO (blood group anti A, anti B antibodies) incompatible donor liver.
4. Patient has fulminant liver failure with a life expectancy without a liver transplant of less than 7 days as defined by UNOS (Adult Patient Status 1, UNOS Policy 3.6.4.1: See Appendix C).
5. Patient has renal dysfunction pre-transplant that, in the opinion of the investigator, will prohibit the use of calcineurin inhibitors within 72 hours post transplant.
6. Patient is intubated, on vasopressors, is ICU bound, or has experienced a significant blood loss (greater than 5 units) 72 hours prior to transplant procedure.
7. Recipient or donor is seropositive for human immunodeficiency virus (HIV) or HbsAg positive serology.
8. Patient is to receive antilymphocyte antibody induction therapy, such as ATGAM (lymphocyte immune globulin), OKT3 (muromonab-CD3), Simulect (basiliximab), or Thymoglobulin.
9. Patient has a known hypersensitivity to Prograf (TAC), HCO-60, CellCept (MMF), Zenapax or corticosteroids.
10. Patient is pregnant or lactating.
11. Patient has participated in a blinded trial or participated in a trial involving a non-marketed (investigational) drug within 3 months of enrollment.
12. Patient has participated in a trial involving a market drug within 30 days. However, patients who participated in any interferon or ribavirin trials are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2002-07; Primary Completion 2006-04 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Goran Klintmalm, MD, Principal Investigator — Baylor Univeristy Medical Center
Locations (1):
- Baylor Regional Transplant Institute - Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No their is not a plan to make individual Participant data available

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period August 15, 2002-March 29, 2004 Recruitment of liver transplant receipeints from centers transplant program
Pre-assignment Details: Subjects must be receiving a liver transplant for end stage chronic HCV
Groups:
- Treatment Arm 1: Immunosuppression TAC (tacrolimus) and CS (cyclosporine)
- Treatment Arm 2: Immunosuppression MMF(mofetil mycophenolate), TAC (tacrolimus) and CS (cyclosporine)
- Treatment Arm 3: Immunosuppression DAC (daclizumub), MMF (mofetil mycophenolate)and TAC (tacrolimus)
Period: Overall Study
Arm/Group | Treatment Arm 1 | Treatment Arm 2 | Treatment Arm 3
Started | 80 | 79 | 153
Completed | 60 | 56 | 116
Not Completed | 20 | 23 | 37
Not completed — Death | 12 | 14 | 19
Not completed — graft loss | 4 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 3 | 2
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Non Compliance | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 10
Not completed — Other reason | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm 1 | Treatment Arm 2 | Treatment Arm 3 | Total
Number analyzed (Participants) | 80 | 79 | 153 | 312
Age, Customized [Mean (Standard Deviation); unit: years]
  Years | 51.7 (7.2) | 51.4 (7.8) | 51.5 (7.4) | 51.6 (7.4)
Gender [Count of Participants; unit: Participants]
  Female | 24 | 19 | 44 | 87
  Male | 56 | 60 | 109 | 225
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80 | 79 | 153 | 312
Reduce HCV recurrent post liver transplant [Number; unit: participants] — Patients receiving a liver transplant for chronic HCV
  participants | 80 | 79 | 153 | 312

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Acute Rejection or HCV Recurrence or Treatment Failure
Description: Freedom from acute rejection (Banff>grade 2 with RAI score>4) or freedom from HCV recurrence (Batts/Ludwig>Stage 2, or >Grade 3) that requires HCV antiviral therapy or treatment failure (patient death, graft loss, premature withdrawal from study regimen or treatment with more than 1 dose of corticosteroids for presumptive rejection without a biopsy to confirm the rejection; reported values represent the "Number of participants with Freedom From Acute Rejection or HCV Recurrence or Treatment Failure"
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Treatment Arm 1 | Treatment Arm 2 | Treatment Arm 3
Number analyzed (Participants) | 80 | 79 | 153
participants | 69 | 70 | 133

2. Primary Outcome: Freedom From HCV Recurrence Within First Year That Requires HCV Antiviral Therapy and Freedom From Treatment Failure
Description: Participants would have their blood drawn and tested for the HCV virus to determine if they had recurrence
Time Frame: 12 month post transplant
Measure: Number; unit: participants
Arm/Group | Treatment Arm 1 | Treatment Arm 2 | Treatment Arm 3
Number analyzed (Participants) | 80 | 79 | 153
participants | 39 | 39 | 72

ADVERSE EVENTS:
Time Frame: 24 months
Description: biopsy, labs
Arm/Group | Treatment Arm 1 | Treatment Arm 2 | Treatment Arm 3
Serious Adverse Events (participants affected / at risk) | 12/80 | 14/79 | 14/153
Other Adverse Events (participants affected / at risk) | 12/80 | 79/79 | 153/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm 1 (N=80) | Treatment Arm 2 (N=79) | Treatment Arm 3 (N=153)
Death (General disorders) | 12 (12) | 14 (14) | 14 (19)
Graft loss (General disorders) | 4 (4) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm 1 (N=80) | Treatment Arm 2 (N=79) | Treatment Arm 3 (N=153)
thrombocytopenia (General disorders) | 5 (6) | 40 (45) | 80 (85)
neutropenia (General disorders) | 3 (4) | 40 (45) | 70 (75)
anemia (General disorders) | 4 (5) | 40 (45) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less